CLINICAL TRIAL: NCT05973734
Title: Clinical Islet Transplantation With Apheresis, Isolation and Reintroduction of Recipient Regulatory T Cells or Administration of Deceased Donor Vertebral Bone Marrow in Type 1 Diabetes
Brief Title: Islet Transplantation With Recipient T-Reg Cells or Deceased Donor Vertebral Bone Marrow Therapy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Stephan Busque, Protocol Director, Stanford University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 58350
Record Dates: First submitted 2023-06-14; First posted 2023-08-03 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Islet Transplantation

STUDY DESIGN:
Intervention Model Description: All patients are planned to receive an islet transplantation. The patients will also receive either Arm 1) recipient T regulatory cell infusion or arm 2) same donor vertebral body derived bone marrow cell infusion. Attribution to either arm will be based on the availability of either cell product in specific cases.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Recipient T Regulatory Cell (Experimental): T regulatory cells prior to islet transplantation, induction therapy with ATG and Belatacept and maintenance immunosuppression with Tacrolimus Extended-release tablets (Envarsus XR) and Mycophenolate Mofetil (MMF).
  Interventions: Biological: Infusion of recipient T regulatory cell
- Donor Derived Vertebral Bone Marrow (Experimental): Deceased donor vertebral bone marrow (VBM) cells, induction therapy with ATG and Belatacept and maintenance immunosuppression with Tacrolimus Extended-release tablets (Envarsus XR) and Mycophenolate Mofetil (MMF).
  Interventions: Biological: Infusion of concomitant Donor Derived Vertebral Bone Marrow

INTERVENTIONS:
Biological: Infusion of recipient T regulatory cell — Patients will undergo a single apheresis collection with a target total blood volume of 20-30 L and the collected cells used as the source of purified Tregs to be infused following the islet transplantation. In the event a patient is unable to meet the collection target, a second collection may be performed.
  Arms: Recipient T Regulatory Cell
Biological: Infusion of concomitant Donor Derived Vertebral Bone Marrow — The cells from the donor VB and spleen are processed under cGMP conditions and released for infusion after the respective recipient has undergone transplant and conditioning. Under this protocol, the donor's VB will be obtained at the same time as the pancreatic islets and will be the source of HSC for infusion with the intent to establish immune tolerance to the donor's pancreatic islet cells. Subjects will receive one infusion of allogeneic cadaveric islets. Subjects will receive induction therapy with ATG and Belatacept and maintenance immunosuppression with Tacrolimus Extended-release tablets (Envarsus XR) and Mycophenolate Mofetil (MMF). After islet transplantation, the VBM cells will be infused in one time window: on day 0-1. Subjects will undergo closed-loop insulin pump glucose control peri-transplant.
  Arms: Donor Derived Vertebral Bone Marrow

SUMMARY:
The goal of this clinical trial is to learn if patients who have brittle type 1 diabetes receiving an islet transplantation will have better control of their sugars if they also receive one of 2 types of immune cells along with the islet transplant. The participants will receive either their own immune cells, called regulatory T cells, or immune cells from the bone marrow of the islet donor.

DETAILED DESCRIPTION:
Islet transplantation success remains limited by the immediate loss of islet after transplantation, rejection, and side effect from immunosuppression. Preclinical animal models provide evidence that donor bone marrow cells OR regulatory T cells infused at the time of islet transplantation can improve the survival of islets after transplantation and reduce the need for immunosuppression. The purpose of this study is to evaluate the feasibility and safety of combining an islet transplant with the recipient's Tregs OR deceased donor bone marrow cells in patients with brittle type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients age 18 to 70 years of age.
* Ability to provide written informed consent.
* Mentally stable and able to comply with the procedures of the study protocol.
* Clinical history compatible with T1D with onset of disease at < 45 years of age, insulin- dependence for ≥ 5 years at the time of enrollment, or a sum of patient age and insulin dependent diabetes duration of ≥ 28.
* Absence of stimulated C peptide (< 0.3 ng/mL) in response to a mixed meal tolerance test measured at 60 and 90 minutes after the start of consumption
* Involvement in intensive diabetes management defined as self-monitoring of glucose values no less than a mean of three times each day averaged over each week and by the administration of three or more insulin injections each day or insulin pump therapy. Such management must be under the direction of an endocrinologist, diabetologist, or diabetes specialist with at least 3 clinical evaluations during the 12 months prior to study enrollment.
* At least two episodes of severe hypoglycemia in the 12 months prior to study enrollment.
* Reduced awareness of hypoglycemia as defined by a Clarke score of 4 or more OR a HYPO score greater than or equal to the 90th percentile (1047) during the screening period and within the last 6 months prior to randomization.
* Women of childbearing potential may be enrolled if a pregnancy test is negative, and they agree to the use of 2 forms of contraception from Screening to the end of the study. Males must agree to use 2 forms of contraception from Screening to the end of the study if their partners are of childbearing potential.
* Acceptable methods of birth control which must be used together are:

  * Oral contraceptive and condom (combination oral contraceptives containing the second- generation progestin (levonorgestrel) and <30 μg of estrogen should be utilized),
  * IUD and condom,
  * Diaphragm with spermicide and condom
* Subject must complete training on how to use the Tandem X2 pump with Control IQ technology by a certified Diabetes Educator or physician. Patients must complete at least 2 hour training to the satisfaction of the educator and show proficiency and understanding in its use as judged by the educator.
* Patients with prior kidney transplantation on immunosuppressive medications are eligible provided they meet all eligibility criteria above excluding the need for hypoglycemia unawareness. Patients should not be candidates for solid organ pancreas transplant or have declined the surgical option.
* Exclusion Criteria:
* Body mass index (BMI) >30 kg/m2 or patient weight ≤50kg.
* Insulin requirement of >1.0 IU/kg/day or <15 U/day. 3. HbA1c >10%.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of Screening
* Untreated proliferative diabetic retinopathy.
* Blood Pressure: SBP >180 mmHg or DBP >100 mmHg on optimal treatment.
* Estimated glomerular filtration rate of <50 mL/min/1.73m2.
* Presence or history of macroalbuminuria (>500mg/g creatinine).
* Presence or history of panel-reactive anti-HLA antibodies >50%. Negative cross- match by flow cytometry and no DSA to organ donor by standard methods.
* For female subjects: Positive pregnancy test, presently breast-feeding, or unwillingness to use effective contraceptive measures for the duration of the study and 4 months after discontinuation. For male participants: intent to procreate during the duration of the study or within 4 months after discontinuation or unwillingness to use effective measures of contraception
* Presence of active infection including hepatitis B, hepatitis C, HIV, or tuberculosis (TB). Subjects with laboratory evidence of active infection are excluded even in the absence of clinical evidence of active infection.
* Negative screen for Epstein-Barr Virus (EBV) by IgG determination.
* Invasive aspergillus, histoplasmosis, or coccidioidomycosis infection within one year prior to study enrollment.
* Any history of malignancy except for completely resected squamous or basal cell carcinoma of the skin.
* Known active alcohol or substance abuse.
* Baseline Hb below the lower limits of normal; neutropenia (<1,500/7L), or thrombocytopenia (platelets <100,000/7L).
* Any coagulopathy or medical condition requiring long-term anticoagulant therapy (e.g., warfarin) after islet transplantation (low-dose aspirin treatment is allowed) or patients with an international normalized ratio (INR) >1.5.
* Severe co-existing cardiac disease, characterized by any one of these conditions:

  * recent myocardial infarction (within past 6 months).
  * evidence of uncorrectable ischemia on functional cardiac exam within the last year.
  * left ventricular ejection fraction <30%.
* Persistent elevation of liver function tests at the time of study entry. Persistent serum glutamic-oxaloacetic transaminase (SGOT [AST]), serum glutamate pyruvate transaminase (SGPT [ALT]), or total bilirubin, with values > 1.5 times normal upper limits will exclude a patient.
* Acute or chronic pancreatitis.
* Treatment with any anti-diabetic medication other than insulin within 4 weeks of enrollment.
* Use of any investigational agents within 4 or more weeks of enrollment, depending upon the pharmacokinetics of the investigational agent and durability of changes with treatment in immune function or glycemic regulation.
* Administration of live attenuated vaccine(s) within 2 months of enrollment.
* Any medical condition that, in the opinion of the investigator, will interfere with safe participation in the trial.
* A previous islet transplant.
* History of medical non-adherence or poor social support.
* Individuals with selective IgA deficiencies (IgA level less than 15 mg/dL) who have known antibody against IgA.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
Occurrence of Grade 3 to 5 cytokine release syndrome / acute infusion reaction after Treg administration infusion reaction after Treg administration | within 3 months
  Grade 3 to 5 cytokine release syndrome / acute infusion reaction after Treg administration infusion reaction after Treg administration
Occurrence of grade 4 or greater adverse events of islet transplantation | Within two years
  Adverse event grade 4 or greater
Number of patients who receive Treg infusions (Arm1) or Donor Derived Vertebral Bone Marrow (Arm2) and islet transplantation (feasibility) | Within two years
  Number of patients who received planned Treg or Donor Bone Marrow

SECONDARY OUTCOMES:
HbA1c ≤6.5% | assessed at 6, 12 and 24 months post-islet transplantation
  HbA1c ≤6.5%
Absence of severe hypoglycemic events | assessed at 6, 12 and 24 months post-islet transplantation
  Absence of severe hypoglycemic event , requiring intervention by other person than the patient
Decrease of insulin mean requirements (u/kg) from prior to transplantation by 50% of total daily dose | assessed at 6, 12 and 24 months post-islet transplantation
  Reduction of exogenous insulin requirement by 50% from baseline
Clarke hypoglycemia severity (HYPO) score less than 2 (0 to >4, >4 indicate severe hypoglycemia unawareness) | assessed at 6, 12 and 24 months post-islet transplantation
  Improvement of Clarke score to less than 2
Basal C-peptide at levels e >0.5 ng/mL (>0.17 nmol/L) fasting or stimulated. | assessed at 6, 12 and 24 months post-islet transplantation
  C-petide production from islet transplant assessment
Target of glucose variability and hypoglycemia duration derived from the CGMS <Standard Deviation and Coefficient targets> | assessed at 6, 12 and 24 months post-islet transplantation
  Monitoring of glucose control 24h sensor monitoring
Measurement of donor Specific Antibody, cPRA | assessed at 6, 12 and 24 months post-islet transplantation
  Single bead luminex anti HLA class 1 and 2 assay
Quality of life (QOL) assessment | assessed at 6, 12 and 24 months post-islet transplantation
  QOL questionnaire SF-12 (0-100, higher score is better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Busque, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ryan EA, Shandro T, Green K, Paty BW, Senior PA, Bigam D, Shapiro AM, Vantyghem MC. Assessment of the severity of hypoglycemia and glycemic lability in type 1 diabetic subjects undergoing islet transplantation. Diabetes. 2004 Apr;53(4):955-62. doi: 10.2337/diabetes.53.4.955. PMID 15047610
- [Background] Kessler L, Passemard R, Oberholzer J, Benhamou PY, Bucher P, Toso C, Meyer P, Penfornis A, Badet L, Wolf P, Colin C, Morel P, Pinget M; GRAGIL Group. Reduction of blood glucose variability in type 1 diabetic patients treated by pancreatic islet transplantation: interest of continuous glucose monitoring. Diabetes Care. 2002 Dec;25(12):2256-62. doi: 10.2337/diacare.25.12.2256. PMID 12453970
- [Background] Streja D. Can continuous glucose monitoring provide objective documentation of hypoglycemia unawareness? Endocr Pract. 2005 Mar-Apr;11(2):83-90. doi: 10.4158/EP.11.2.83. PMID 15901522
- [Background] Diabetes Control and Complications Trial Research Group; Nathan DM, Genuth S, Lachin J, Cleary P, Crofford O, Davis M, Rand L, Siebert C. The effect of intensive treatment of diabetes on the development and progression of long-term complications in insulin-dependent diabetes mellitus. N Engl J Med. 1993 Sep 30;329(14):977-86. doi: 10.1056/NEJM199309303291401. PMID 8366922
- [Background] Hirsch IB. Insulin analogues. N Engl J Med. 2005 Jan 13;352(2):174-83. doi: 10.1056/NEJMra040832. No abstract available. PMID 15647580
- [Background] Cryer PE, Davis SN, Shamoon H. Hypoglycemia in diabetes. Diabetes Care. 2003 Jun;26(6):1902-12. doi: 10.2337/diacare.26.6.1902. PMID 12766131
- [Background] Gold AE, MacLeod KM, Frier BM. Frequency of severe hypoglycemia in patients with type I diabetes with impaired awareness of hypoglycemia. Diabetes Care. 1994 Jul;17(7):697-703. doi: 10.2337/diacare.17.7.697. PMID 7924780
- [Background] Larsen JL. Pancreas transplantation: indications and consequences. Endocr Rev. 2004 Dec;25(6):919-46. doi: 10.1210/er.2002-0036. PMID 15583023
- [Background] Cryer PE, Fisher JN, Shamoon H. Hypoglycemia. Diabetes Care. 1994 Jul;17(7):734-55. doi: 10.2337/diacare.17.7.734. No abstract available. PMID 7924788
- [Background] Ryan EA, Paty BW, Senior PA, Bigam D, Alfadhli E, Kneteman NM, Lakey JR, Shapiro AM. Five-year follow-up after clinical islet transplantation. Diabetes. 2005 Jul;54(7):2060-9. doi: 10.2337/diabetes.54.7.2060. PMID 15983207
- [Background] Hering BJ, Clarke WR, Bridges ND, Eggerman TL, Alejandro R, Bellin MD, Chaloner K, Czarniecki CW, Goldstein JS, Hunsicker LG, Kaufman DB, Korsgren O, Larsen CP, Luo X, Markmann JF, Naji A, Oberholzer J, Posselt AM, Rickels MR, Ricordi C, Robien MA, Senior PA, Shapiro AM, Stock PG, Turgeon NA; Clinical Islet Transplantation Consortium. Phase 3 Trial of Transplantation of Human Islets in Type 1 Diabetes Complicated by Severe Hypoglycemia. Diabetes Care. 2016 Jul;39(7):1230-40. doi: 10.2337/dc15-1988. Epub 2016 Apr 18. PMID 27208344
- [Background] Krzystyniak A, Golab K, Witkowski P, Trzonkowski P. Islet cell transplant and the incorporation of Tregs. Curr Opin Organ Transplant. 2014 Dec;19(6):610-5. doi: 10.1097/MOT.0000000000000130. PMID 25304813
- [Background] Pierini A, Iliopoulou BP, Peiris H, Perez-Cruz M, Baker J, Hsu K, Gu X, Zheng PP, Erkers T, Tang SW, Strober W, Alvarez M, Ring A, Velardi A, Negrin RS, Kim SK, Meyer EH. T cells expressing chimeric antigen receptor promote immune tolerance. JCI Insight. 2017 Oct 19;2(20):e92865. doi: 10.1172/jci.insight.92865. PMID 29046484
- [Background] Cryer PE. Banting Lecture. Hypoglycemia: the limiting factor in the management of IDDM. Diabetes. 1994 Nov;43(11):1378-89. doi: 10.2337/diab.43.11.1378. PMID 7926315
- [Background] Shapiro AM, Lakey JR, Ryan EA, Korbutt GS, Toth E, Warnock GL, Kneteman NM, Rajotte RV. Islet transplantation in seven patients with type 1 diabetes mellitus using a glucocorticoid-free immunosuppressive regimen. N Engl J Med. 2000 Jul 27;343(4):230-8. doi: 10.1056/NEJM200007273430401. PMID 10911004
- [Background] Markmann JF, Deng S, Huang X, Desai NM, Velidedeoglu EH, Lui C, Frank A, Markmann E, Palanjian M, Brayman K, Wolf B, Bell E, Vitamaniuk M, Doliba N, Matschinsky F, Barker CF, Naji A. Insulin independence following isolated islet transplantation and single islet infusions. Ann Surg. 2003 Jun;237(6):741-9; discussion 749-50. doi: 10.1097/01.SLA.0000072110.93780.52. PMID 12796569
- [Background] Meyer EH, Laport G, Xie BJ, MacDonald K, Heydari K, Sahaf B, Tang SW, Baker J, Armstrong R, Tate K, Tadisco C, Arai S, Johnston L, Lowsky R, Muffly L, Rezvani AR, Shizuru J, Weng WK, Sheehan K, Miklos D, Negrin RS. Transplantation of donor grafts with defined ratio of conventional and regulatory T cells in HLA-matched recipients. JCI Insight. 2019 May 16;4(10):e127244. doi: 10.1172/jci.insight.127244. eCollection 2019 May 16. PMID 31092732
- [Background] Huber BC, Ransohoff JD, Ransohoff KJ, Riegler J, Ebert A, Kodo K, Gong Y, Sanchez-Freire V, Dey D, Kooreman NG, Diecke S, Zhang WY, Odegaard J, Hu S, Gold JD, Robbins RC, Wu JC. Costimulation-adhesion blockade is superior to cyclosporine A and prednisone immunosuppressive therapy for preventing rejection of differentiated human embryonic stem cells following transplantation. Stem Cells. 2013 Nov;31(11):2354-63. doi: 10.1002/stem.1501. PMID 24038578
- [Background] Bellacen K, Kalay N, Ozeri E, Shahaf G, Lewis EC. Revascularization of pancreatic islet allografts is enhanced by alpha-1-antitrypsin under anti-inflammatory conditions. Cell Transplant. 2013;22(11):2119-33. doi: 10.3727/096368912X657701. Epub 2012 Oct 8. PMID 23050776
- [Background] Hubbard RC, Sellers S, Czerski D, Stephens L, Crystal RG. Biochemical efficacy and safety of monthly augmentation therapy for alpha 1-antitrypsin deficiency. JAMA. 1988 Sep 2;260(9):1259-64. PMID 3261353
- [Background] Baranovski BM, Ozeri E, Shahaf G, Ochayon DE, Schuster R, Bahar N, Kalay N, Cal P, Mizrahi MI, Nisim O, Strauss P, Schenker E, Lewis EC. Exploration of alpha1-antitrypsin treatment protocol for islet transplantation: dosing plan and route of administration. J Pharmacol Exp Ther. 2016 Dec;359(3):482-490. doi: 10.1124/jpet.116.236067. Epub 2016 Nov 7. PMID 27821710
- [Background] Weir GC, Ehlers MR, Harris KM, Kanaparthi S, Long A, Phippard D, Weiner LJ, Jepson B, McNamara JG, Koulmanda M, Strom TB; ITN RETAIN Study Team. Alpha-1 antitrypsin treatment of new-onset type 1 diabetes: An open-label, phase I clinical trial (RETAIN) to assess safety and pharmacokinetics. Pediatr Diabetes. 2018 Aug;19(5):945-954. doi: 10.1111/pedi.12660. Epub 2018 May 7. PMID 29473705
- [Background] Koulmanda M, Bhasin M, Fan Z, Hanidziar D, Goel N, Putheti P, Movahedi B, Libermann TA, Strom TB. Alpha 1-antitrypsin reduces inflammation and enhances mouse pancreatic islet transplant survival. Proc Natl Acad Sci U S A. 2012 Sep 18;109(38):15443-8. doi: 10.1073/pnas.1018366109. Epub 2012 Sep 4. PMID 22949661
- [Background] Wang J, Sun Z, Gou W, Adams DB, Cui W, Morgan KA, Strange C, Wang H. alpha-1 Antitrypsin Enhances Islet Engraftment by Suppression of Instant Blood-Mediated Inflammatory Reaction. Diabetes. 2017 Apr;66(4):970-980. doi: 10.2337/db16-1036. Epub 2017 Jan 9. PMID 28069642
- [Background] Berger M, Liu M, Uknis ME, Koulmanda M. Alpha-1-antitrypsin in cell and organ transplantation. Am J Transplant. 2018 Jul;18(7):1589-1595. doi: 10.1111/ajt.14756. Epub 2018 Apr 24. PMID 29607607
- [Background] Taylor GD, Kirkland T, Lakey J, Rajotte R, Warnock GL. Bacteremia due to transplantation of contaminated cryopreserved pancreatic islets. Cell Transplant. 1994 Jan-Feb;3(1):103-6. doi: 10.1177/096368979400300114. PMID 8162286
- [Background] Lloveras J, Farney AC, Sutherland DE, Wahoff D, Field J, Gores PF. Significance of contaminated islet preparations in clinical islet transplantation. Transplant Proc. 1994 Apr;26(2):579-80. No abstract available. PMID 8171564
- [Background] Rickels MR, Kamoun M, Kearns J, Markmann JF, Naji A. Evidence for allograft rejection in an islet transplant recipient and effect on beta-cell secretory capacity. J Clin Endocrinol Metab. 2007 Jul;92(7):2410-4. doi: 10.1210/jc.2007-0172. Epub 2007 May 8. PMID 17488791
- [Background] Rickels MR, Kearns J, Markmann E, Palanjian M, Markmann JF, Naji A, Kamoun M. HLA sensitization in islet transplantation. Clin Transpl. 2006:413-20. PMID 18365398
- [Background] Olack BJ, Swanson CJ, Flavin KS, Phelan D, Brennan DC, White NH, Lacy PE, Scharp DW, Poindexter N, Mohanakumar T. Sensitization to HLA antigens in islet recipients with failing transplants. Transplant Proc. 1997 Jun;29(4):2268-9. doi: 10.1016/s0041-1345(97)00327-8. No abstract available. PMID 9193621
- [Background] Mao Q, Terasaki PI, Cai J, Briley K, Catrou P, Haisch C, Rebellato L. Extremely high association between appearance of HLA antibodies and failure of kidney grafts in a five-year longitudinal study. Am J Transplant. 2007 Apr;7(4):864-71. doi: 10.1111/j.1600-6143.2006.01711.x. PMID 17391129
- [Background] Terasaki PI, Ozawa M. Predicting kidney graft failure by HLA antibodies: a prospective trial. Am J Transplant. 2004 Mar;4(3):438-43. doi: 10.1111/j.1600-6143.2004.00360.x. PMID 14961999
- [Background] Terasaki PI, Ozawa M, Castro R. Four-year follow-up of a prospective trial of HLA and MICA antibodies on kidney graft survival. Am J Transplant. 2007 Feb;7(2):408-15. doi: 10.1111/j.1600-6143.2006.01644.x. Epub 2007 Jan 4. PMID 17229080
- [Background] Epidemiology of severe hypoglycemia in the diabetes control and complications trial. The DCCT Research Group. Am J Med. 1991 Apr;90(4):450-9. PMID 2012085
- [Background] Ramsay RC, Goetz FC, Sutherland DE, Mauer SM, Robison LL, Cantrill HL, Knobloch WH, Najarian JS. Progression of diabetic retinopathy after pancreas transplantation for insulin-dependent diabetes mellitus. N Engl J Med. 1988 Jan 28;318(4):208-14. doi: 10.1056/NEJM198801283180403. PMID 3275895
- [Background] Hirshberg B, Rother KI, Digon BJ 3rd, Lee J, Gaglia JL, Hines K, Read EJ, Chang R, Wood BJ, Harlan DM. Benefits and risks of solitary islet transplantation for type 1 diabetes using steroid-sparing immunosuppression: the National Institutes of Health experience. Diabetes Care. 2003 Dec;26(12):3288-95. doi: 10.2337/diacare.26.12.3288. PMID 14633816
- [Background] Ryan EA, Lakey JR, Paty BW, Imes S, Korbutt GS, Kneteman NM, Bigam D, Rajotte RV, Shapiro AM. Successful islet transplantation: continued insulin reserve provides long-term glycemic control. Diabetes. 2002 Jul;51(7):2148-57. doi: 10.2337/diabetes.51.7.2148. PMID 12086945
- [Background] Ryan EA, Paty BW, Senior PA, Shapiro AM. Risks and side effects of islet transplantation. Curr Diab Rep. 2004 Aug;4(4):304-9. doi: 10.1007/s11892-004-0083-8. PMID 15265474
- [Background] Froud T, Yrizarry JM, Alejandro R, Ricordi C. Use of D-STAT to prevent bleeding following percutaneous transhepatic intraportal islet transplantation. Cell Transplant. 2004;13(1):55-9. doi: 10.3727/000000004772664897. PMID 15040605
- [Background] Hering BJ, Kandaswamy R, Ansite JD, Eckman PM, Nakano M, Sawada T, Matsumoto I, Ihm SH, Zhang HJ, Parkey J, Hunter DW, Sutherland DE. Single-donor, marginal-dose islet transplantation in patients with type 1 diabetes. JAMA. 2005 Feb 16;293(7):830-5. doi: 10.1001/jama.293.7.830. PMID 15713772
- [Background] Manciu N, Beebe DS, Tran P, Gruessner R, Sutherland DE, Belani KG. Total pancreatectomy with islet cell autotransplantation: anesthetic implications. J Clin Anesth. 1999 Nov;11(7):576-82. doi: 10.1016/s0952-8180(99)00100-2. PMID 10624643
- [Background] Froberg MK, Leone JP, Jessurun J, Sutherland DE. Fatal disseminated intravascular coagulation after autologous islet transplantation. Hum Pathol. 1997 Nov;28(11):1295-8. doi: 10.1016/s0046-8177(97)90204-5. PMID 9385936
- [Background] Mehigan DG, Bell WR, Zuidema GD, Eggleston JC, Cameron JL. Disseminated intravascular coagulation and portal hypertension following pancreatic islet autotransplantation. Ann Surg. 1980 Mar;191(3):287-93. doi: 10.1097/00000658-198003000-00006. PMID 6767451
- [Background] Mittal VK, Toledo-Pereyra LH, Sharma M, Ramaswamy K, Puri VK, Cortez JA, Gordon D. Acute portal hypertension and disseminated intravascular coagulation following pancreatic islet autotransplantation after subtotal pancreatectomy. Transplantation. 1981 Apr;31(4):302-4. No abstract available. PMID 6784295